CLINICAL TRIAL: NCT06089278
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trials to Assess the Effectiveness, Safety and Pharmacokinetics of TQH2722 Injection in Patients With Chronic Sinusitis With or Without Nasal Polyps.
Brief Title: A Clinical Study of TQH2722 Injection in the Treatment of Chronic Sinusitis With or Without Nasal Polyps.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2722-II-02
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-04

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 300mg of TQH2722 injection (Experimental): TQH2722 injection, 14 days as a treatment cycle.
  Interventions: Drug: 300mg of TQH2722 injection
- 600mg of TQH2722 injection (Experimental): TQH2722 injection, 14 days as a treatment cycle.
  Interventions: Drug: 600mg of TQH2722 injection
- TQH2722 injection matching placebo (Placebo Comparator): TQH2722 injection matching placebo, 14 days as a treatment cycle.
  Interventions: Drug: TQH2722 injection matching placebo

INTERVENTIONS:
Drug: 300mg of TQH2722 injection — TQH2722 injection is a fully human monoclonal antibody that interfering with the signal cascade.
  Arms: 300mg of TQH2722 injection
Drug: 600mg of TQH2722 injection — TQH2722 injection is a fully human monoclonal antibody that interfering with the signal cascade.
  Arms: 600mg of TQH2722 injection
Drug: TQH2722 injection matching placebo — Placebo without active substance.
  Arms: TQH2722 injection matching placebo

SUMMARY:
To evaluate the effectiveness, safety and pharmacokinetics of TQH2722 injection in patients with chronic sinusitis with or without nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, gender is not limited;
* Bilateral chronic sinusitis (with or without nasal polyps) that meets the diagnostic criteria of The Chinese Guidelines for the Diagnosis and Treatment of Chronic Sinusitis (2018);
* Systemic corticosteroids (at least 1 course of prednisone 0.5 to 1 mg/kg/day or equivalent for at least 5 days) within 2 years prior to the screening, but bilateral chronic sinusitis still exist; and/or patients with drug contraindications/intolerance to systemic glucocorticoids, and (or) patients who have undergone sinus surgery within 6 months before the screening;
* Before the screening, subjects must have used a stable dose of intranasal corticosteroids (INCS) for more than 4 weeks; For participants who used INCS alternatives rather than Mometasone furoate nasal spray (MFNS) prior to screening, participants should be willing to switch to MFNS in the duration of the study;
* Subjects with asthma started inhaled glucocorticoids at a stable dose at least 4 weeks before the screening and could remain inhaled glucocorticoid doses unchanged throughout the study;
* Patients in the Run-in period should be willing to conduct diary, daily symptom assessment and maintain a stable dose of MFNS with at least 70% adherence;
* Be able to read and understand, and be willing to sign informed consent;
* Participants and their partners agreed to use effective contraception throughout the study period (from the beginning of the screening/run-in period to 3 months after the last dose).

Exclusion Criteria:

* Any disease that the investigator considers unstable and may affect the patient's safety throughout the study period, or affect or interpretation with the results, or interfere with the patient's ability to complete the entire research process, including but not limited to cardiovascular, gastrointestinal, liver, kidney, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic diseases, psychiatric disorders, or major limb disorders. For example, but not limited to: ischemic heart disease, left ventricular failure, arrhythmia, uncontrolled hypertension, uncontrolled hyperglycemia, cerebrovascular disease, etc.;
* Patients with active autoimmune disease;
* Known or suspected immunosuppressed, including but not limited to invasive opportunistic infections
* Subjects with active malignant tumors or a history of malignant tumors;
* History of active pulmonary tuberculosis within the 12 months before screening;
* Active hepatitis during the screening period, or positive hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody (HBcAb) and positive hepatitis B virus (HBV) DNA, or positive hepatitis C virus (HCV) antibody and positive HCV-RNA; or positive for antibodies to human immunodeficiency virus (Anti-HIV) or positive for treponemal antibodies (Anti-TP);
* Diagnosed with helminth parasitic infection within 6 months before the screening period, did not receive standard treatment or the standard treatment was ineffective;
* Patients with combined asthma should be excluded if they have:

  1. Forced expiratory volume in the first second (FEV1) ≤ 50% of normal estimates, or
  2. Acute exacerbation of asthma within 90 days prior to screening, requiring hospitalization (>24 hours), or
  3. used daily doses higher than 1000 mcg of fluticasone or equivalent inhaled corticosteroids (ICS);
* The subject had concomitant diseases that prevented him/her from completing the screening period assessment or from evaluating the primary efficacy endpoint;
* Subjects with nasal malignancies and benign tumors (e.g., papillomas, hemangiomas, etc.);
* Subjects who are unable to use MFNS or who are allergic or intolerant to mometasone furoate nasal spray;
* Subjects with a history of anaphylaxis to any biological agent (other than local injection site reactions);
* Pregnant or lactating women;
* Alcoholism, drug addiction and known drug dependence;
* Have participated in clinical trials of other medical devices within 12 weeks before screening;
* The subject had poor compliance in the research and could not complete the study as judged by the investigator;
* In the judgment of the investigator or sponsoring medical reviewer, it is believed that there are any medical or psychiatric symptoms that put the subject at risk, interfere with participation in the study, or interfere with the interpretation of the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in nasal polyp score in Part A | Up to 16 weeks.
  Changes in nasal polyp score in subjects with chronic sinusitis with nasal polyps (CRSwNP) from baseline. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Changes in sinus CT scan Lund Mackay score in Part B | Up to 16 weeks.
  Changes in sinus CT scan Lund Mackay score in subjects with chronic sinusitis without nasal polyps (CRSsNP) from baseline in Part B. The total score is 0-24 points, with the higher score meaning the more severe symptoms.

SECONDARY OUTCOMES:
Changes in sinus CT scan Lund Mackay score in Part A | Up to 16 weeks.
  Changes in sinus CT scan Lund Mackay score in subjects with chronic sinusitis without nasal polyps (CRSsNP) from baseline in Part A. The total score is 0-24 points, with the higher score meaning the more severe symptoms.
Changes in the Lund-Kennedy score by nasal endoscopy | Up to 16 weeks.
  Changes in subjects' nasal endoscopy modified Lund-Kennedy score from baseline. The total score is 0-20 points, with the higher score meaning the more severe symptoms.
Changes in University of Pennsylvania Smell Identification Test (UPSIT) | Up to 16 weeks.
  Changes in University of Pennsylvania Smell Identification Test (UPSIT) of patients from baseline. The total score is 0-40 points, with the lower score meaning the more severe symptoms.
Changes in Nasal Total Symptom Score (sTSS) | Up to 16 weeks.
  Changes in subjects' Nasal Total Symptom Score (sTSS) from baseline. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Changes in the Anosmia score | Up to 16 weeks.
  Changes in subjects' Anosmia scores from baseline. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in nasal congestion score (NCS) | Up to 16 weeks.
  Change in subjects' Nasal congestion Score (NCS) from baseline at week 16. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in nasal/post-nasal discharge scores | Up to 16 weeks.
  Changes in subjects' nasal/post-nasal discharge scores from baseline at week 16. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in facial pain/pressure scores | Up to 16 weeks.
  Changes in subjects' facial pain/pressure scores from baseline. The total score is 0-3 points, with the higher score meaning the more severe symptoms.
Changes in the Visual analogue Scale (VAS) of sinusitis | Up to 16 weeks.
  Changes in the Visual Analogue Scale (VAS) for sinusitis in subjects from baseline. The total score is 0-10 points, with the higher score meaning the more severe symptoms.
Subjects' Health-related Quality of Life (HRQoL) questionnaire | Up to 16 weeks.
  Effects of Subjects' Health-related Quality of Life (HRQoL) from baseline. The total score is 0-100 points, with the higher score meaning the more severe symptoms.
Changes in nasal peak inspiratory flow rate (NPIF) | Up to 16 weeks.
  Changes in the subject's nasal peak inspiratory flow rate (NPIF) from baseline
Systemic glucocorticoid (SCS) remedial or surgical treatment rate | Up to 16 weeks.
  Proportion of patients receiving systemic glucocorticoid (SCS) remedial or surgical treatment during 16 weeks
Incidence of adverse events | Up to 24 weeks.
  Incidence of adverse events (AES) and serious adverse events (SAEs), as well as abnormal laboratory test indicators
Severity of adverse events | Up to 24 weeks.
  Severity of adverse events (AES) and serious adverse events (SAEs), as well as abnormal laboratory test indicators
Peak concentration (Cmax) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  Maximum plasma drug concentration
Trough concentration (Cmin) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  Minimum plasma drug concentration
Peak time (Tmax) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The time required to reach peak concentration after administration
Area under blood concentration-time curve (AUC0-t) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The area enclosed by the blood concentration curve to the timeline
Steady-state peak concentration (Css-max) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The highest blood concentration that occurs in steady state
Steady-state valley concentration (Css-min) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The lowest blood concentration that occurs in steady state
Mean steady-state blood concentration (Css-av) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The quotient obtained by dividing the area under the blood concentration-time curve by the interval time τ during a dose interval when the blood concentration reaches a steady state
Steady-state peak time (Tss-max) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The time required to reach peak steady-state concentration after administration
Area under steady state blood concentration-time curve (AUC ss,0-t) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  Area under the blood concentration-time curve in steady state
Elimination half-life | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The time it takes for half the drug to be eliminated from the body
Apparent volume of distribution (Vd/F) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  The ratio of the amount of drug in the body to the concentration in the blood after the drug has reached homeostasis in the body
Clearance rate (CL/F) | Within 1 hour before and 1, 4, 8, 12, 24, 72, 168 hours after the first dose; Within 1 hour before the 2nd, 3rd, and 6th doses; Within 1 hour before and 1, 4, 8, 12, 24, 48, 72, 168, 336, 672, 840 hours after the last dose.
  Per unit time, the volume of drug-containing liquid is completely and effectively removed by the elimination organ

CONTACTS AND LOCATIONS:
Locations (36):
- China (36):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing TongRen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Foshan First People's Hospital, Foshan, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated hospital of Guizhou Medical University, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospitalc, Tongji Medical College, Huazhong, University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Loudi Central Hospital, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The Affiliated Hospital of Yanbian University, Yanji, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Shandong Second People's Hospital, Jinan, Shandong
  - Weifang Second People's Hospital, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Wenling First People's Hospital, Taizhou, Zhejiang
  - Taizhou central hospital, Taizhou, Zhejiang